CLINICAL TRIAL: NCT00806832
Title: The Effects of Medical Clowning on Blood Pressure and Pulse Rate of Patients Undergoing Cataract Surgery Under Local Anesthesia
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Yaron Lang, MD, Department of Ophthalmology, HaEmek MC, Afula, Israel
Other Study IDs: 0087-08-EMC
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Blood Pressure; Heart Rate
Keywords: Medical clowns; Cataract surgery; Blood pressure; Heart rate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Medical clowns treatment: Patients scheduled for an elective cataract surgery will receive pre-operative conventional treatment and in addition will be exposed to medical clowns effect
- Conventional treatment only: Patients scheduled for elective cataract surgery will receive only conventional pre-operative treatment

SUMMARY:
Cataract surgery is the most prevalent surgical procedure. Since most candidates are elderly patients, hypertension is common among these patients. Preoperative anxiety and tension may cause elevation of patient's heart rate and blood pressure and thus expose them to serious potential complications such as stroke and myocardial infarction. Medical clowns are known to reduce preoperative anxiety of both children and their parents. It is possible therefore that medical clown may have such a beneficial effect also on patients scheduled for cataract surgery under local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective, ambulatory cataract surgery (phacoemulsification technique)
* Surgery planned to be performed under local anesthesia
* Age > 40 years
* Patients signed an informed consent

Exclusion Criteria:

* Hypertensive patients who did not take their prescribed medications on the day of surgery
* Uncontrolled hypertension during the month preceding the surgery
* Patients with systolic and diastolic BP values of >190 and 100 mmHg respectively, measured 1hr prior to surgery
* Patients not suitable for surgery under local anesthesia
* Patients in whom the planned phacoemulsification technique was converted to either the ECCE or ICCE technique
* Patients in whom an anterior vitrectomy had to be performed during surgery
* Patients treated regularly by anti-anxiety or analgetic treatment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients from the town of Afula and its surrounding region who are scheduled for cataract surgery in Ha'Emek Medical Center.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Blood pressure | day of surgery

SECONDARY OUTCOMES:
heart rate | day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Lang, MD, Principal Investigator — Dept. of Ophthalmology, Ha'Emek MC, Afula, Israel
Locations (1):
- Department of Ophthalmology, Ha'Emek MC, Afula, Israel

REFERENCES:
- [Background] Vagnoli L, Caprilli S, Robiglio A, Messeri A. Clown doctors as a treatment for preoperative anxiety in children: a randomized, prospective study. Pediatrics. 2005 Oct;116(4):e563-7. doi: 10.1542/peds.2005-0466. PMID 16199685